CLINICAL TRIAL: NCT06526845
Title: Examining The Effectiveness of Telerehabilitation in Individuals With Temporomandibular Joint Dysfunction and Myofascial Pain
Brief Title: Effectiveness of Telerehabilitation in Individuals With Temporomandibular Joint Dysfunction and Myofascial Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Collaborators: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Buket AKINCI, Assoc. Prof., Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-54022451-050.04-144681
Record Dates: First submitted 2024-07-17; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Temporomandibular Joint Dysfunction; Myofascial Pain
Keywords: Temporomandibular Joint Disorders; Telerehabilitation; Exercise
MeSH Terms: conditions — Temporomandibular Joint Disorders; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation Group (Experimental): All exercises in the brochure will be performed by patients via telerehabilitation.It will be applied twice a week for 6 weeks.
  Interventions: Other: Video-Conference based rehabilitation
- Home-Based Exercise Group (Active Comparator): Patient education will be provided by showing all the exercises in practice. Then, brochures will be given to the patients so that they can practice them at home.It will be applied twice a week for 6 weeks.
  Interventions: Other: Home-Based rehabilitation

INTERVENTIONS:
Other: Video-Conference based rehabilitation — All exercises in the brochure will be performed by patients via telerehabilitation. The exercises included in the exercise package are as follows:
  * Post-isometric relaxation exercise and relaxation exercise with diaphragmatic breathing
  * Neck Exercises: 5 neck exercises including cervical isometric flexion, extension, right and left lateral flexion and chin tuck exercises.
  * Soft tissue-friction massage: It will be applied to the area where myofascial pain develops due to TMJD.
  * Mandibular mobility exercises: opening and closing the mouth slowly and rhythmically, lateral movements, protrusion movement, hold-relax technique, jaw isometric exercises
  * Stretching exercises: Stretching exercises for chewing muscles (masseter muscle stretching, temporalis muscle stretching, pterygoid muscle stretching).
  Arms: Telerehabilitation Group
Other: Home-Based rehabilitation — Patient education will be provided by showing all exercises in practice. Brochures will then be given to patients so they can apply them at home. The exercises in the brochure are as follows;
  * Post-isometric relaxation exercise and relaxation exercise with diaphragmatic breathing
  * Neck Exercises: 5 neck exercises including cervical isometric flexion, extension, right and left lateral flexion and chin tuck exercises.
  * Soft tissue-friction massage: It will be applied to the area where myofascial pain develops due to TMJD.
  * Mandibular mobility exercises: opening and closing the mouth slowly and rhythmically, lateral movements, protrusion movement, hold-relax technique, jaw isometric exercises
  * Stretching exercises: Stretching exercises for chewing muscles (masseter muscle stretching, temporalis muscle stretching, pterygoid muscle stretching).
  Arms: Home-Based Exercise Group

SUMMARY:
Telerehabilitation is a treatment method that allows the patient to access treatment remotely, regardless of where they are, thanks to developing technology. Telerehabilitation provides us with opportunities such as patient evaluation, monitoring, therapy, consultation, education and patient follow-up. Within the scope of our study, the effects of applying an exercise program to patients through a home exercise program and telerehabilitation will be investigated. The purpose of this study for individuals with temporomandibular joint dysfunction is; To investigate the effectiveness of exercises for myofascial pain through telerehabilitation in individuals with myofascial pain and TMJ dysfunction.

DETAILED DESCRIPTION:
TMJ, one of the most complex joints of the body, is a ginglimoarthrodial joint located in the front part of the external auditory canal, between the mandibular fossa (glenoid fossa) of the temporal bone and the condylar processes of the mandible, and also performs rotation and sliding movements. It is composed of fibrous connective tissue between the bone tissues that form the joint. There is a joint disc that divides the joint space into two parts, lower and upper. TMJ is effective in basic functions such as providing mandibular movement, speaking and chewing. A normal person uses TMJ a lot in daily life. For this reason, pathologies related to TMJ are encountered more frequently than other joints in the body. Clinical signs and symptoms of temporomandibular joint disorders may vary, but pain, noise from the joint, limitation of mandibular movements and tenderness in the chewing muscles are among the most frequently observed symptoms. It has been shown in many studies that the daily living activities of individuals with TMJ dysfunction are negatively affected, and this affects the quality of life of individuals. Therefore, identification, diagnosis and treatment of symptoms are important. Many methods such as analgesic and anti-inflammatory drugs, splint therapy, exercise and physical therapy modalities are used in the treatment of these individuals. When looking at the literature, it is seen that exercise therapy has an important place in TMJ rehabilitation and that a supervised rehabilitation program is effective in improving functional parameters. In the studies of Çapan et al., it was seen that active exercise and relaxation exercises applied to the chewing muscle groups were an effective treatment method on deviation and pain. Bae et al. showed that manual therapy and exercise applications for the cervical region had positive effects on pain threshold in chewing muscles and pain-free mouth opening in patients with myofascial type TMD. In a systematic review published in 2014, joint mobilization, soft tissue mobilization and friction massage were recommended to reduce pain, increase normal joint movement (ROM) and reduce other symptoms within the scope of manual therapy techniques (MTT) for TMJ problems. Especially in soft tissue mobilization, the method called pressure trigger point release technique; It is a noninvasive method based on gradually applying pressure on the trigger point in accordance with the patient's tolerance. Exercise is one of the approaches that have been used for a long time in the treatment of TMJ problems. Therapeutic exercises specific to TMJ problems can be used to specifically improve the functions between the TMJ and the craniomandibular system. Most exercise programs have an important place in increasing muscle coordination, normalizing range of motion, providing muscle relaxation and increasing muscle strength.

Telerehabilitation is a treatment method that allows the patient to access treatment remotely, regardless of where they are, thanks to developing technology. Telerehabilitation provides us with opportunities such as patient evaluation, monitoring, therapy, consultation, education and patient follow-up. Within the scope of our study, the effects of applying an exercise program to patients through home exercise program and telerehabilitation will be investigated.

The purpose of this study for individuals with temporomandibular joint dysfunction; To investigate the effectiveness of exercises for myofascial pain through telerehabilitation in individuals with myofascial pain and TMJ dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* People between the ages of 18-65 with myofascial temporomandibular pain
* Displacement of the disc with anterior reduction,
* Pain in the masticatory muscle/temporomandibular area lasting more than a month
* Symptoms lasting at least three months,
* People who have the opportunity to provide informed consent and participate in treatment and evaluation clinics.

Exclusion Criteria:

* Anterior disc displacement without reduction,
* Primary arthrogenic pain,
* Other temporomandibular disorders,
* Neurological or psychiatric disorders,
* People who have had temporomandibular joint and/or cervical spine surgery,
* Abuse of painkillers or abuse of existing medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-23 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Fonseca Anamnestic Index | Change from Fonseca Anamnestic Index at 6 weeks.
  Temporomandibular dysfunction is assessed using the Fonseca Anamnestic Index .
Visual Analogue Scale | Change from Visual Analog Scale at 6 weeks.
  Participants; It is performed to evaluate jaw and facial pain when waking up in the morning, during the day, at bedtime, when chewing and at rest.
  Visual Analogue Scale includes scoring between 0-10. The minimum value is 0 score - no pain; The maximum score of 10 indicates unbearable pain. A higher score means more pain and a worse outcome.
Painless Maximum Mouth Opening | Change from Painless Maximum Mouth Opening at 6 weeks.
  It will be done to evaluate the painless maximum mouth opening of the participants.
  It will be performed to evaluate the pain-free maximum mouth opening of the participants.
  The patient will be asked to open his mouth as far as possible and the distance between the lower and upper incisors will be measured with a millimeter ruler. The result will be recorded in mm.
Painful Maximum Mouth Opening | Change from Painful Maximum Mouth Opening at 6 weeks.
  It will be performed to evaluate the participants' maximum mouth opening with pain.
  The patient will be asked to open his mouth to the last painful point and the distance between the lower and upper incisors will be measured with a millimeter ruler. The result will be recorded in mm.
Maximum Mouth Opening With Passive Assistance | Change from Maximum Mouth Opening With Passive Assistance at 6 weeks.
  It will be carried out to evaluate the maximum mouth opening of the participants with passive assistance (dentist or physiotherapist).
  The patient will be asked to open his mouth as far as possible with the support of a dentist or physiotherapist, and the distance between the lower and upper incisors will be measured with a millimeter ruler. The result will be recorded in mm.
Mandibula Lateral Shift | Change from Mandibula Lateral Shift at 6 weeks.
  It evaluates the right and left shifts of the mandibula in participants. The patient first moves his lower jaw to the right and how far it moves from the midline is measured with a millimetric ruler. The measured value is recorded in millimeters. Then, the same process is performed for the left side.
Oral Health Impact Profile-14 (OHIP-14) | Change from Oral Health Impact Profile-14 (OHIP-14) at 6 weeks.
  It evaluates the quality of life in temporomandibular joint dysfunction. The total score varies between 0-84. A high score indicates that you have bad oral habits.

SECONDARY OUTCOMES:
Oral Behaviour Checklist | Change from Oral Behaviour Checklist at 6 weeks.
  It is applied to evaluate the oral behaviour of the participants.
Cervical Region Joint Range of Motion | Change from Cervical Region Joint Range of Motion at 6 weeks.
  It will be applied to evaluate the participants cervical region flexion, extension, right and left lateral flexion, and right and left rotation degrees.
Neck Disability Index | Change from Neck Disability Index at 6 weeks.
  The NDI measures self-reported pain intensity (pain, headache) and limitations in performing daily work-related activities (work, lifting and concentration) and non-work-related activities (personal care, reading, driving, sleeping and leisure).

CONTACTS AND LOCATIONS:
Overall Officials: Buket AKINCI, Assoc.Prof., Study Director — Consultor; Nükhet KÜTÜK, Prof., Study Chair — study chair; Beliz SERDAROĞLU, Dt., Study Chair — study chair; Naile FAZLIOĞLU, PT., Principal Investigator — Study Principal Investigator
Locations (1):
- Buket AKINCI, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The data will be shared during the publication process if the journal will ask.